CLINICAL TRIAL: NCT03254732
Title: Phase 1B Study of ADI-PEG 20 Plus Pembrolizumab in Advanced Solid Cancers
Brief Title: Study ADI-PEG 20 Plus Pembrolizumab in Advanced Solid Cancers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Changing Corporate Priorities
Sponsor: Polaris Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POLARIS2016-002
Record Dates: First submitted 2016-12-23; First posted 2017-08-18 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2020-03

CONDITIONS: Advanced Solid Cancers
MeSH Terms: interventions — ADI PEG20; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ADI-PEG 20 (Experimental): This is a phase 1b, open label trial of ADI-PEG 20 (36 mg/m2) weekly in combination with pembrolizumab (1 and 2 mg/kg or 200 mg) every three weeks.
  Interventions: Drug: ADI PEG20; Drug: Pembrolizumab

INTERVENTIONS:
Drug: ADI PEG20 — ADI is a recombinant protein cloned from M. hominis and produced in E. coli, and conjugated with PEG of 20,000 mw. Thus ADI-PEG 20 is an arginine degrading enzyme, ADI, coupled to PEG.
Drug: Pembrolizumab — Pembrolizumab is a PD-1 blocking antibody indicated in the USA for the treatment.
  Other Names: Keytruda®

SUMMARY:
This is a phase 1b, open label trial of ADI-PEG 20 (36 mg/m2) weekly in combination with pembrolizumab (1 and 2 mg/kg or 200 mg) every three weeks. Assessment of safety and tolerability of drug combination

DETAILED DESCRIPTION:
This is an open-label, phase 1b trial of ADI-PEG 20 in combination with pembrolizumab in subjects with advanced cancers. Dose escalation will occur using a 3 + 3 + 3 design.

The first subject in a dose escalation cohort must have had treatment with ADI-PEG 20 + pembrolizumab with a week of follow up) before the next 2 subjects are enrolled. Thus subjects 2 and 3 may be enrolled on day 8 if there is no dose limiting toxicity (DLT) in subject 1. No additional delay is required between treating subjects 4 to 6 or 7 to 9 in an expanded cohort. Before proceeding to the next cohort dose level, the first 3 eligible subjects in each cohort will have received at least 21 days of treatment (i.e. at least 2 of the expected 3 doses of ADI-PEG 20 + one dose of pembrolizumab).

ELIGIBILITY:
Select Inclusion Criteria:

1. Histologically confirmed diagnosis of advanced solid tumor.
2. Prior failure of a systemic treatment approved by the health authority in the country where the study will be enrolling. Such subjects may also have been treated with radiotherapy, local therapy or surgery.
3. Measurable disease using RECIST 1.1 criteria.
4. Age ≥ 18 years.

Select Exclusion Criteria:

1. Subjects with history of another primary cancer, including co-existent second malignancy, with the exception of: a) curatively resected non-melanoma skin cancer; b) curatively treated cervical carcinoma in situ; or c) other primary solid tumor with no known active disease present or in the opinion of the investigator will not affect patient outcome.
2. Subjects who had been treated with ADI-PEG 20 previously.
3. History of seizure disorder not related to underlying cancer.
4. Known allergy to pegylated compounds.
5. Known allergy to E. coli drug products (such as GMCSF).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-07-14 (Actual); Primary Completion 2019-05-07 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability of ADI-PEG 20 in combination with Pembrolizumab in Advanced Solid Cancers | Up to 36 months
  Number of participants with treatment-related adverse events and severity this is graded by CTCAE and MedDRA for Coding

SECONDARY OUTCOMES:
Number of Participants with PFS with Combination ADI-PEG 20 and Pembro. | Assessments ever 9 weeks for 12 months
  Progression Free Survival determined by RECIST 1.1
Number of Participants with RR with Combination ADI-PEG 20 and Pembro. | Assessments ever 9 weeks for 12 months
  Response Rate determined by RECIST 1.1

OTHER OUTCOMES:
Overall Survival | 12 months after end of treatment
  Follow-Up by Phone or Clinic Visit

CONTACTS AND LOCATIONS:
Locations (1):
- Facility National Cheng Kung University, Tainan, Taiwan